CLINICAL TRIAL: NCT00115089
Title: A Phase II Multi-Center, Randomized, Double-Blind, Active and Placebo-Controlled 7 Day Study of Mast Cell Inhibitor, R926112, in Patients With Symptomatic Seasonal Allergic Rhinitis
Brief Title: 7 Day Study of Mast Cell Inhibitor, R926112, in Patients With Symptomatic Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-926112-005A
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Last update posted 2005-11-11 (Estimated); Status verified 2005-11

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Allergic Rhinitis; Nasal Spray; Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — Beclomethasone

INTERVENTIONS:
Drug: R926112
Drug: Beclomethasone dipropionate

SUMMARY:
This is a study of the effectiveness and safety of a new nasal spray for the relief of the symptoms of seasonal allergies. The agents being compared are: R926112 (a novel anti-allergy medicine), Beconase (beclomethasone dipropionate, an established FDA approved steroid treatment), and an inactive placebo. The study hypothesis is that R926112 will be superior to placebo at the end of a week of testing and evaluation. The study does not have the power to determine how R926112 compares to Beconase.

DETAILED DESCRIPTION:
Seven hundred fifty patients with histories of seasonal allergies will be screened in late summer and early fall at 25 sites across the U.S. Approximately 375 patients, based on severity of symptoms will be randomized among the treatments (150 to R926112, 150 to placebo, 75 to Beconase). During, and for about 2-3 weeks prior to the study, patients will have to abstain from other anti-allergy medications. Patients will fill out diary cards two times per day to record their symptoms. The entire study should take between 2-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign a written informed consent form and assent (if applicable) for study participation.
* Males and females, 12 years of age or older
* Subjects must have a history consistent with seasonal allergic rhinitis (SAR) during the fall pollen season for at least the previous 2 years.
* Subjects must be skin test positive to a relevant fall aeroallergen within the past 12 months with at least a moderate reaction as defined by at least a 5 mm wheal.
* Nasal exam to exclude significant swelling, bleeding, crusting, or polyps
* Subjects receiving immunotherapy must be on a stable maintenance regimen for at least 30 days before screening. Adjustments to the regimen following a brief period of missed injections or the normal reduction in dose due to a vaccine refill does not preclude participation.
* Female subjects of childbearing potential must have negative urine tests for pregnancy at Visits 1 and 2.
* Female subjects of childbearing potential who are sexually active will be expected to use a medically recognized birth control method throughout the study: systemic contraceptive (oral, implant, injection, patch), diaphragm with intravaginal spermicide, cervical cap, vaginal ring, intrauterine device, or condom with spermicide. Females who are not sexually active will be admitted by the discretion of the Investigator. Acceptable birth control will be documented in the subject's case report form.
* Subjects must be willing to adhere to dosing schedules, study visits, and study requirements.

Exclusion Criteria:

* Clinically significant medical conditions (such as hepatic, neurological, hematological, renal, cardiac, gastrointestinal, endocrine, or other major systemic disease), which in the judgment of the Investigator, might interfere with the study, require treatment or make implementation of the protocol or interpretation of the study results difficult.
* Clinically relevant abnormalities in laboratory results or electrocardiogram (ECG) as determined by the investigator
* Asthma that requires treatment other than with inhaled, short acting beta agonist alone.
* Female subjects who are pregnant, trying to become pregnant, or nursing.
* Nasal structural abnormalities, including large nasal polyps or marked septal deviation that significantly interfere with nasal airflow or nasal surgery within the past year.
* Upper respiratory infection within 3 weeks before the date of Randomization/Visit 2.
* Treatment with any investigational drug in the last 30 days before the date of Randomization/Visit 2.
* History of drug or alcohol abuse that according to the Investigator could interfere with the study.
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
* Subjects unlikely to comply with study procedures, unable to return for study visits, or unlikely to complete the study, or expecting or planning to travel outside the area of the prevalent aeroallergen during the study period.
* History of hypersensitivity to steroids or to the excipients.
* Use of tricyclic antidepressants within the past 30 days prior to date of Randomization/Visit 2.
* Ocular herpes simplex or cataracts present at the time of Screening Visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 375
Dates: Start 2005-07; Study Completion 2005-09

PRIMARY OUTCOMES:
Change in total nasal symptom score from baseline over time

SECONDARY OUTCOMES:
Change in individual symptoms
Global therapeutic response
Quality of life score

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Grossbard, M.D., Study Director — Rigel Pharmaceuticals; Eli Meltzer, M.D., Principal Investigator — Allergy and Asthma Medical Group and Research Center, San Diego; Harold Nelson, M.D., Principal Investigator — National Jewish Medical Research Center, Denver

REFERENCES:
- [Background] Meltzer EO, Berkowitz RB, Grossbard EB. An intranasal Syk-kinase inhibitor (R112) improves the symptoms of seasonal allergic rhinitis in a park environment. J Allergy Clin Immunol. 2005 Apr;115(4):791-6. doi: 10.1016/j.jaci.2005.01.040. PMID 15806000